CLINICAL TRIAL: NCT00000270
Title: Brain Imaging: Cocaine Effects & Medication Development
Brief Title: Brain Imaging: Cocaine Effects & Medication Development - 5
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never opened; never enrolled participants
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-09236-5; 5P50DA009236-18 (NIH); P50-09236-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cocaine

SUMMARY:
The purpose of this study is to define temporal profile of brain activation (rCBF) using Xenon-SPECT and O 15-PET.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1995-12-30 (Actual); Primary Completion 1995-12-30 (Actual); Study Completion 1995-12-30 (Actual)

PRIMARY OUTCOMES:
Absolute change in rCBF at 5 & 15 minutes (Xe)
Relative change in rCBF at 5, 19, & 33 minutes (O15)
Correlated with a) subjective effects, b) venous blood level of coca, c) autonomic variables

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] ACNP Abstract, 1995. CPDD Abstract, 1996. Society for Nuclear Medicine, 1996. Society for Neuroscience, 1997.